CLINICAL TRIAL: NCT06544187
Title: Can Imaging be an Alternative to Exercise Testing as a Predictor of Surgical Fitness?
Acronym: RESPIRE
Status: Recruiting | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 3354
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Surgical Fitness; Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants: The first phase of the study will involve 56 participants who are potential candidates for oesophagectomy, gastrectomy or pancreaticoduodenectomy procedures following a confirmed cancer diagnosis. Participants who provide their consent will undergo Magnetic Resonance Spectroscopy (MRS) scans of their semitendinosus muscle in the thigh. Participants on this pathway also undergo Cardiopulmonary Exercise Test (CPET) tests, which is a standard procedure. No delay to their normal treatment pathway will be introduced from the addition of the MRS scan, and MR scans can be arranged within two weeks from referral
  Interventions: Diagnostic Test: MRS scan; Diagnostic Test: CPET
- Healthy volunteers: 25 healthy volunteers. Their role will be to help us understand the consistency in Intra-Myocellular Liquid (IMCL) composition using Magnetic Resonance Spectroscopy (MRS) techniques. These volunteers will be sourced from the UHNM Trust staff, in accordance with Trust Standard Operating Procedure (SOP): The Safe Scanning of Volunteers in Magnetic Resonance Imagine (MRI). Each volunteer will undergo two MRS scans initially. All three MRS scans will be performed in a single session, with the session lasting about 20 minutes. Additionally, each volunteer will return for a single repeat session of MRS acquisition using the same MRI system and protocol, scheduled at two weeks after the initial scans
  Interventions: Diagnostic Test: MRS scan; Diagnostic Test: CPET

INTERVENTIONS:
Diagnostic Test: MRS scan — Magnetic Resonance Spectroscopy scan on the thigh
Diagnostic Test: CPET — Cardiopulmonary Exercise Test

SUMMARY:
This study aims to explore an alternative method for assessing a participant's readiness for surgery, specifically for those undergoing surgery for gastric, oesophageal, or pancreatic cancer. Surgery for these diseases is extremely demanding on the body and surgeons need to be confident that a patient can tolerate the procedure.

Traditionally, participants undergo Cardiopulmonary Exercise Tests (CPET) to determine their fitness for surgery. This involves cycling on an exercise bike with increasing resistance until the resistance is too great to continue cycling at a constant rate. An individual's maximum rate of oxygen consumption (VO2max) and the anaerobic threshold (AT) are calculated during CPET and used by surgeons as a predictor for surgical fitness. CPET tests can be physically demanding for participants and are very resource intensive. Furthermore, some patients may not be able to tolerate exercise tests due to physical constraints.

An alternative method, Magnetic Resonance Spectroscopy (MRS), could be used to measure an individual's fitness prior to surgery. Within this study, MRS will be used to determine the levels of fat within the thigh muscle, which in turn may be able to be used to predict fitness for surgery.

The first phase includes recruiting participants on the surgical pathway. MRS will be performed as an additional examination, typically on the same day as the CPET. Fat levels determined from MRS will be compared with conventional CPET outcomes (VO2max and AT). This analysis aims to determine if MRS derived fat levels correlates with VO2max and AT and, if correlation is high, potentially providing an alternative to CPET for patients who cannot tolerate exercise tests.

The second phase involves recruiting volunteers who will undergo repeated MRS scans to assess the reliability of MRS methods. This process allows us to understand the consistency of MRS derived fat levels over both short and long-term intervals.

The potential benefits of this project include an additional pathway for assessing fitness for surgery or enhancing the presurgical pathway for patients by providing an alternative method for fitness assessment. This study aims to provide evidence that could present an alternative method of assessing a patient's fitness for surgery. The goal is to explore an alternative that may complement or refine current practices in preoperative assessments.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients (cohort 1)

* Patients diagnosed oesophageal/gastric or pancreatic cancer.
* Patients who have or a under consideration for a CPET investigation.
* Aged ≥ 18.
* Existing UHNM Patient.
* Willing and able to give fully informed consent.
* Willing and able to comply with the study procedures.

Inclusion criteria for staff volunteers (cohort 2)

* Aged ≥ 18 years.
* Willing and able to give fully informed consent.
* Willing and able to comply with the study procedures.
* UHNM member of staff.

Exclusion Criteria:

Exclusion criteria for patients (cohort 1)

* Patients with contraindications to MRI due to safety at 3T.
* Patients with metalwork within the imaging field of view (e.g., knee replacement).
* Claustrophobic patients.
* Patients outside of stated age range to ensure informed consent.
* Patients not referred for CPET investigations.
* Patients that are pregnant.
* Patients that are unable to communicate in English.
* Patients lacking the capacity and capability to give fully informed consent.
* Patients participating in any other interventional studies with a contraindication to their participation.
* Patients for whom the addition of an MRS scan would delay any part of their standard treatment pathway.
* History of diabetes.

Exclusion criteria for staff volunteers (cohort 2)

* Volunteers with contraindications to MRI due to safety at 3T.
* Volunteers with metalwork within the imaging field of view (e.g., knee replacement).
* Claustrophobic volunteers.
* Volunteers outside of stated age range to ensure informed consent.
* Volunteers that are pregnant.
* Volunteers that are unable to communicate in English.
* Volunteers lacking the capacity and capability to give fully informed consent.
* Volunteers participating in any other interventional studies with a contraindication to their participation.
* Known or suspected medical conditions pertinent to the area being scanned.
* History of diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1: Participants with oesophageal, gastric or pancreatic cancer who are potential candidates for surgical resection (oesophagectomy/gastrectomy/pancreaticoduodenectomy).
  Cohort 2: Healthy volunteers who are UHNM staff members ≥ 18 years old, with no known contraindication to MRI. Volunteers will be age and gender matched to the participants in cohort 1.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Correlations between levels | 2 years
  Calculate the correlation between the intramyocellular lipid (IMCL) saturation index and Cardiopulmonary Exercise Test (CPET) derived VO2max and Anaerobic Threshold (AT).

SECONDARY OUTCOMES:
Comparisons between participants who did not suffer major morbidity | 2 years
  Compare the mean Intra-Myocellular Lipid (IMCL) saturation index for patients who suffered major morbidity after oesophagectomy, gastrectomy, or pancreaticoduodenectomy and compare this to the mean IMCL saturation index of those who did not suffer major morbidity.
Short and long term repeatability | 2 years
  Assess the short- and long-term repeatability of Magnetic Resonance Spectroscopy (MRS) of Intra-Myocellular Lipid (IMCL) saturation index measurements in healthy volunteers.
  .
Difference in IMCL composition | 2 years
  Assess the difference in Intra-Myocellular Lipid (IMCL) composition between patients considered for surgery and age and gender matched volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared